CLINICAL TRIAL: NCT03133078
Title: Impact of Fatigue on Jumping Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 959318
Record Dates: First submitted 2016-11-17; First posted 2017-04-28 (Actual); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Healthy
Keywords: Side Hop; Forward Hop; Step test; Vertical Jump

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise: step-down test (2 min) (Experimental): The 2-minute single limb lateral-step down test will be used to induce lower extremity muscle fatigue. Participants will be instructed to perform a single limb lateral step-down test on a 31 cm box (12-inches), touching their heel to the floor each time as many times as possible in 2 minutes. The number of lateral step-downs will be recorded.
  Interventions: Other: Step-Down Test (2 min)
- Exercise: side hop test (30 s) (Experimental): The 30 second side hop test will be used to induce lower extremity muscle fatigue. Participants will be instructed to jump as many times as possible over two parallel strips of tape placed 40 cm apart, but must initiate approximately 30 degrees of knee flexion each jump. The number of successful jumps performed within 30 seconds will be recorded and used for data analysis. An unsuccessful jump will be defined as touching the tape or the area inside the tape. We will record the number of successful trials.
  Interventions: Other: Side hop test (30 s)

INTERVENTIONS:
Other: Step-Down Test (2 min) — The 2-minute single limb lateral-step down test will be used to induce lower extremity muscle fatigue. Participants will be instructed to perform a single limb lateral step-down test on a 31 cm box (12-inches), touching their heel to the floor each time as many times as possible in 2 minutes. The number of lateral step-downs will be recorded.
  Arms: Exercise: step-down test (2 min)
Other: Side hop test (30 s) — The 30 second side hop test will be used to induce lower extremity muscle fatigue. Participants will be instructed to jump as many times as possible over two parallel strips of tape placed 40 cm apart, but must initiate approximately 30 degrees of knee flexion each jump. The number of successful jumps performed within 30 seconds will be recorded and used for data analysis. An unsuccessful jump will be defined as touching the tape or the area inside the tape. We will record the number of successful trials.
  Arms: Exercise: side hop test (30 s)

SUMMARY:
The purpose of this study will be to determine the effects of a 2-minute single limb lateral step-down fatigue test versus a 30 second side hop test on single limb forward hop distance.

DETAILED DESCRIPTION:
Current methods to induce fatigue often incorporate equipment not available in all clinical settings or include tasks that are difficult to standardize. One of the tests to fatigue the leg muscles is the leg extensor fatigue test using a unilateral weight machine. There are drawbacks to this testing including the clinician having access to the equipment, testing only fatigued a single muscle group, and it is less sport/task specific compared to jump testing. Our previous work has incorporated the use of a side hop task that is performed by hopping over two lines 40 cm apart for 30 seconds. While this does induce fatigue and decreases single leg forward hop performance the overall decrease was relatively small (<10 cm). It is likely necessary to induce a greater amount of fatigue; thus further limiting single leg forward hop performance.

ELIGIBILITY:
Inclusion Criteria:

* No history of knee surgery
* Tegner score >5

Exclusion Criteria:

* Participants with traumatic spine or lower extremity injury within past 6 months
* Participants who are unable to give consent or are unable to understand procedures of experiment

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-11; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Single limb hop distance (cm) | Change from baseline single limb hop distance immediately after fatigue exercise
  While standing on one leg participants will be instructed to hop as far forward as possible with a controlled single limb landing.

CONTACTS AND LOCATIONS:
Overall Officials: Terry L Grindstaff, PhD, PT, ATC, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No